CLINICAL TRIAL: NCT03832283
Title: Patient Outcomes Reporting for Timely Assessments of Life With Depression: PORTAL-Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QI18-90
Record Dates: First submitted 2019-02-01; First posted 2019-02-06 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Depression; Depressive Disorder, Major
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Masking Description: Patients randomized to MyChart will not be blinded to the intervention. Patients who are randomized to usual screening will not be informed about the intervention arm and, thus, will be blinded to trial assignment. PCPs will not be informed of the randomization; however, they will receive results whenever their patients complete the CAT-MH via MyChart.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care Depression Screening (Other): Patients randomized to this intervention arm will receive usual care annual depression screening when they come in for a clinic visit and are due for screening. When the patient comes in for a visit, a best practice alert in the EHR will indicate that the patient requires depression screening. The CAD-MDD/CAT-DI screening during clinic visit will occur in a patient room, prior to their appointment with a primary care provider.
  Interventions: Diagnostic Test: CAD-MDD/CAT-DI screening during clinic visit
- Population MyChart Depression Screening (Experimental): Patients randomized to this intervention arm will continue to receive usual care annual depression screening when they come in for a clinic visit and are due for screening. In addition, they will receive email invitations to complete the CAD-MDD/CAT-DI screening via MyChart. Email invitations will be sent at preset intervals until depression screening is completed, or the end of the 1-year follow-up period, whichever comes first.
  Interventions: Diagnostic Test: CAD-MDD/CAT-DI screening via MyChart; Diagnostic Test: CAD-MDD/CAT-DI screening during clinic visit
- Usual Care Depression Monitoring (Other): Patients who have depression and are randomized to this intervention arm will receive usual care PHQ-9 monitoring during clinic visits. When the patient comes in for a visit, a best practice alert in the EHR will indicate that the patient requires depression assessment.
  Interventions: Other: PHQ-9 monitoring during clinic visits
- Population MyChart Depression Monitoring (Experimental): Patients who have depression and are randomized to this intervention arm will continue to receive usual care depression monitoring when they come for clinic visits. In addition, they will receive email invitations at preset intervals to complete the CAT-DI monitoring via MyChart. Invitations will be sent until major depressive disorder (MDD) remission is achieved, or the 1-year follow-up period ends, whichever comes first.
  Interventions: Other: CAT-DI monitoring via MyChart; Other: PHQ-9 monitoring during clinic visits

INTERVENTIONS:
Diagnostic Test: CAD-MDD/CAT-DI screening via MyChart — Patients will receive invitations via MyChart to complete the CAD-MDD to screen for major depressive disorder (MDD). For patients who screen positive for MDD, CAT-DI will launch automatically and assess depression severity. CAT-DI assigns a score of 0 to 100 in four severity categories (<50=normal, 50 to 65=mild, 66 to 75=moderate, and >75=severe).
  Arms: Population MyChart Depression Screening
Diagnostic Test: CAD-MDD/CAT-DI screening during clinic visit — During routine in-clinic visits, medical assistants or providers will ask patients to complete the CAD-MDD to screen for major depressive disorder (MDD). For patients who screen positive for MDD, CAT-DI will launch automatically and assess depression severity. CAT-DI assigns a score of 0 to 100 in four severity categories (<50=normal, 50 to 65=mild, 66 to 75=moderate, and >75=severe).
  Arms: Population MyChart Depression Screening; Usual Care Depression Screening
Other: CAT-DI monitoring via MyChart — Patients with active MDD will receive invitations via MyChart to complete the CAT-DI to assess MDD severity and remission. A normal CAT-DI score (<50) will indicate that a patient's MDD is in remission.
  Arms: Population MyChart Depression Monitoring
Other: PHQ-9 monitoring during clinic visits — During routine in-clinic visits, medical assistants or providers will ask patients to complete the PHQ-9 to assess MDD severity and remission. A PHQ-9 score < 5 will indicate that a patient's MDD is in remission.
  Arms: Population MyChart Depression Monitoring; Usual Care Depression Monitoring

SUMMARY:
Currently, very little research exists on whether patient portals could be used to integrate patient-reported outcome (PRO) measurement into the electronic health record (EHR) and clinical practice, even though 87% of ambulatory care practices have EHRs and 88% of U.S. adults have access to the internet. To date, no randomized controlled trial has examined whether patient portals can be used to collect PRO measures. The goal of this study is to implement the integration of a computerized adaptive test (CAT) for patient-reported outcome (PRO) measurement of depression symptoms into an electronic health record (EHR) and evaluate the effectiveness of collecting CAT PROs via an EHR patient portal in two randomized controlled trials. This study will advance the science of implementation of patient-centered outcomes research into clinical practice, as well as the evidence for high quality, accessible care.

DETAILED DESCRIPTION:
The overall goal of this proposal is to implement the integration of the Computerized Adaptive Test for Mental Health (CAT-MH) into an EHR for a healthcare system and evaluate the effectiveness of collecting CAT-MH PROs via an EHR-tethered patient portal (MyChart) vs. usual care in two randomized controlled trials. The first aim of this study will consist of a randomized controlled trial comparing screening rates among adult primary care patients with an active patient portal account (MyChart) and due for depression screening who receive usual care (CAT-MH screenings during routine clinic visits) vs. MyChart population-based CAT-MH screenings. The second aim of this study involves a randomized controlled trial comparing depression remission rates among patients with active moderate-to-severe MDD who receive usual care vs. MyChart CAT-MH measurement-based care. In addition, we will examine the resources needed to integrate the CAT-MH into the EHR and design the health IT strategy for collecting PROs via the patient portal.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* considered an active clinic patient at the start date of the intervention
* have an active MyChart account that is not managed by a proxy
* receive care from a participating PCP
* due for depression screening (screening arms) or active depression (monitoring arms)

Exclusion Criteria:

* under 18 years of age
* bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4161 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients screened for depression using the BPA by study arm | 12 months
Percentage of patients who have MDD remission | 12 months
Time to MDD remission | 12 months

SECONDARY OUTCOMES:
Percentage of logins to MyChart in response to the email invitations | 12 months
Percentage of opened MyChart depression screening messages | 12 months
Number of MyChart messages sent to PCPs by patients (or to patients by PCPs) following depression screening | 12 months
Percentage of patients who start the CAT-MH assessment | 12 months
Percentage of patients who complete the CAT-MH assessment | 12 months
Percentage of positive screens | 12 months
Number of appointments scheduled and completed (primary care and psychiatry/psychology) | 12 months
Number of telephone encounters in the week following the positive depression screen | 12 months
Number of emergency department visits or hospitalizations due to MDD | 12 months
Percentage of logins to MyChart in response to MyChart emails | 12 months
Percentage of opened MyChart depression symptom measurement messages | 12 months
Number of MyChart messages sent to PCPs by patients (or to patients by PCPs) following completion of the CAT-DI | 12 months
Percentage of patients who start CAT-DI assessments | 12 months
Depression severity scores (CAT-DI) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Staab EM, Franco MI, Zhu M, Wan W, Gibbons RD, Vinci LM, Beckman N, Yohanna D, Laiteerapong N. Population Health Management Approach to Depression Symptom Monitoring in Primary Care via Patient Portal: A Randomized Controlled Trial. Am J Med Qual. 2023 Jul-Aug 01;38(4):188-195. doi: 10.1097/JMQ.0000000000000126. Epub 2023 Jun 15. PMID 37314235
- [Derived] Franco MI, Staab EM, Zhu M, Knitter A, Wan W, Gibbons R, Vinci L, Shah S, Yohanna D, Beckman N, Laiteerapong N. Pragmatic Clinical Trial of Population Health, Portal-Based Depression Screening: the PORTAL-Depression Study. J Gen Intern Med. 2023 Mar;38(4):857-864. doi: 10.1007/s11606-022-07779-9. Epub 2022 Sep 20. PMID 36127535